CLINICAL TRIAL: NCT03043859
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of the Pure Prairie Living Program - A Lifestyle Intervention
Brief Title: A Trial to Evaluate the Effectiveness of the Pure Prairie Living Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Sherwood Park Strathcona County Primary Care Network, Alberta (Unknown)
Responsible Party: Principal Investigator, Catherine Chan, Professor, Dept. of Agriculture Food and Nutritional Sciences, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00070736
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled trial of two arms [intervention (PPLP) and wait-listed controls (CON)]. Baseline data will be collected from all participants. PPLP participants will then receive 5 educational session on healthy eating, behaviour change and lifestyle in addition to usual care, whereas the controls will only receive usual care (no education intervention). Data for primary outcomes will be collected at 3 and 6 month period (from baseline). After the 6 month assessment all participants from the Control group will then recieve intervention and will complete the 3 and 6 month assessments.
Who Masked: Participant, Investigator
Masking Description: Participants who have consented to participate in this study will be assigned a number, those who receive an even number will be assigned to the intervention arm and those who receive an odd number will be in the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pure Prairie Living Program (Experimental): Participants in the intervention arm will participate in 5 weekly education sessions ( 2hours / session) on nutrition education and healthy lifestyle.
  Interventions: Behavioral: Pure Prairie Living Program
- Wait Listed Control (No Intervention): Participants in the control arm will not receive any intervention.

INTERVENTIONS:
Behavioral: Pure Prairie Living Program — Education session (n=5) on healthy eating, menu planning and skill building for effective diabetes management
  Arms: Pure Prairie Living Program

SUMMARY:
In Canada, there is a growing burden of type 2 diabetes (T2D). Approaches to implement nutrition recommendations and promote sustainable eating behaviours are required. The investigating research team developed an educational curriculum that includes practical information about Eating Well with Canada's Food Guide, portion control and food label reading. The research team also developed a cookbook, "Pure Prairie Eating Plan" which translates the Canadian Diabetes Association Clinical Practice Guidelines into a practical menu plan with recipes, grocery lists and cooking tips. These resources promote behaviour change and skill development to independently manage diabetes. These resources have been successfully employed in a clinical study trial conducted at the University of Alberta and in a pilot project at the community (Pure Prairie Living Program -PPLP), and showed beneficial effects in management of diabetes among participants. The objective of this study is to implement and evaluate the PPLP in a community level, to promote healthy lifestyle among people with T2D in the general community. To meet the study objective, 60 adult participants with diagnosed T2D will be recruited from three different primary care networks (total of 180 participants) and at each site 30 participants will be randomized into the education intervention (PPLP) and 30 will be the wait-listed controls (CON) receiving usual care. PPLP participants will attend 5, biweekly education sessions and a grocery store tour scheduled over a period of 3 months.The benefits of the lifestyle intervention on physiological indicators (BMI, Haemoglobin A1C, blood lipids, blood pressure) and lifestyle choices (adherence to dietary recommendations, self-efficacy and participation in physical activity) will be examined.

DETAILED DESCRIPTION:
Overall Goal: To implement and evaluate the effectiveness of a lifestyle intervention (LI) tailored to Albertans' environment called the Pure Prairie Living Program (PPLP) in primary care network (PCN) settings. The PPLP delivers innovation in the concept (based on the 4-A Framework), the setting (PCNs) and nutrition evaluation tools (for Dietary Adherence - PDAQ).

Background: In Canada, there is a growing burden of type 2 diabetes (T2D). One in four Canadians has diabetes or pre-diabetes and this number is projected to be 1 in 3 by 2020. The associated economic burden is estimated to be $16.9 billion in 2020.

Adopting a healthy lifestyle can prevent and also help effectively manage T2D. Several dietary LI in the recent decades have targeted achieving a healthy body weight, participation in physical activity, and healthy eating as primary goals of their intervention trials to delay the progression of the disease or to minimize co-morbidities associated with T2D. Although some of the programs have achieved success in improving health outcomes and delaying the risk of co-morbidities, sustaining long-term changes by the participants after completion of intervention trials is challenging.

Many interventions attempt to personalize treatment based on an individual's preferences and circumstances but fewer consider individual factors within a broader framework of health determinants that includes local food Availability, financially/physically Accessibility, culturally Acceptability and nutritionally Adequacy (4A Framework). Failure to achieve long-term adherence may be influenced by these social and environmental health determinants. Further, Healthcare Professionals (HCP) are designated with the primary responsibility of educating patients to prevent, treat and manage chronic diseases. However HCPs often lack the training, skills, confidence, and time required to implement effective LI and primary care delivery models often lack the required structure and organization for such LI. Few studies consider the health care system-level changes that are required to offer sustainable, high quality LI or programs. Hence to achieve sustained adoption and maintenance of the effects of a LI at a system level requires careful planning (considering the barriers for change, ongoing support to personnel and participants, adopting a framework for behaviour change, improving self-efficacy), implementation and evaluation of the interventions.

In Alberta, Primary Care Networks (PCNs) were implemented to provide citizens access to a multi-disciplinary care team of clinicians, including dietitians. One of the goals of PCNs is to increase the emphasis on health promotion, disease and injury prevention, and care of patients with complex problems or chronic disease. Therefore, the PCN setting is ideal for implementation of LI. The investigators will use the RE-AIM (Reach, Effectiveness, Adoption, Implementation and Maintenance) framework in planning and evaluating the PPLP.

Previous Work by the Research Team: The investigating research team (1) created and validated a simple, practical instrument for assessing dietary adherence to Canadian Diabetes Association (CDA) guidelines called Perceived Dietary Adherence Questionnaire (PDAQ). 2) created and published a 4-week menu plan and recipe book (Pure Prairie Eating Plan, PPEP) to promote healthy eating in the general population and in those with diabetes (www.pureprairie.ca). The menus provide 28 days of suggestions for meeting recommendations of Eating Well with Canada's Food Guide (EWCFG) and CDA nutrition therapy guidelines and incorporate the principles of the 4-A Framework; 3)Pilot tested the menu plan/recipes in 15 participants with T2D and observed a 1.0% reduction in haemoglobin A1C (HbA1c) (p<0.05) after 3 months, along with significant reduction in weight and increase in PDAQ score; 4) In a research setting conducted a single-arm phase 2 trial with 73 volunteer participants with T2D. HbA1c was reduced by 0.7% (p<0.05). Improvements in PDAQ score, serum lipids, blood pressure and self-efficacy were also observed. 5) Based on the successful phase 2 trial, the investigators collaborated with the Southside PCN in Edmonton to pilot an education program centered around PPEP in a patient population. At the system level to ensure suitability of the program, PCN and research personnel refined the education program incorporating information and resources that the PCN was using in existing programming while highlighting the key messages of the education program developed from the phase 2 trial. The program was called PPLP and was piloted in 26 individuals. At an individual level, preliminary results from 17 participants show significantly increased PDAQ score and diabetes self-efficacy along with weight loss.

Specific Objectives: (1) To evaluate the efficacy of PPLP in promoting better nutrition choices (as recommended by EWCFG and CDA Nutrition Therapy Guidelines), improved diabetes self-efficacy, participation in physical activity and improved health outcomes (improved glucose control, lipid panel and blood pressure); (2) To describe the perceived strengths, limitations, effectiveness and satisfaction of the PPLP by HCP and study participants.

Methods:

Study Design: This is a randomized, controlled trial (RCT) of two arms [intervention (PPLP) and wait-listed controls (CON)]. Evaluation will utilize the RE-AIM Framework using mixed methods.

Study Sites: Study will be implemented at 3 PCNs in Edmonton. Site personnel will be co-investigators in the research to facilitate maximal buy-in and integrated knowledge translation (KT). Prior to implementation of the study, the research personnel will offer support to PCN team to develop site specific PPLP protocol and provide necessary training.

Sample Size and Recruitment: A convenience sampling procedure will be employed to recruit study participants through advertisement and posters at the participating PCNs. Investigators aim to recruit a total of 180 participants, 60 participants from each site (30 participants in each RCT arm). Inclusion criteria are: adults (aged 30-80 years) with T2D and able to read and write in English. Exclusion criteria are: having severe gastrointestinal issues or diabetes complications requiring specialized diet or type 1 diabetes.

Procedure

Objective 1) To evaluate the efficacy of PPLP: This intervention study will span 6 months from recruitment to the final participant visit. Details of each visit are as follows:

1. Baseline Assessment (Clinic Visit 1): Weight and height will be measured to calculate body mass index (BMI). Body composition will be assessed using Bio-impedance analyser. Questionnaires to assess demographic information, diabetes management, diabetes self-efficacy, dietary intake pattern (PDAQ), quality of life and physical activity will be completed by participants. Blood pressure (BP) will be assessed and blood sampled for Hb A1C and lipid profile tests. Physical activity will be quantitatively assessed by using pedometers for 3 days. All the data will be collected by a Registered nurse/Dietitian at the PCN. Patients will then be randomized to PPLP or CON groups who will receive usual care prior to enrolment in the intervention.
2. Implementation of the Intervention (Clinic Visit 2-7): PPLP participants will attend and participate in 5, biweekly nutrition and physical activity education sessions (~ 90 min each) that will be conducted at the PCNs' facilities and facilitated by the PCN dietitian. Participants will also be taken for a grocery store tour.
3. 3 Month Assessment (Visit 8): All PPLP and CON participants will visit the PCN, and complete all the questionnaires, blood tests and measurements that were done at Visit 1.
4. Follow-up: All participants will be contacted via phone follow-up on 2 occasions (once a month) to answer any questions related to nutrition and physical activity.
5. 6 Month Assessment (Clinic Visit 9): All PPLP and CON participants will return to the PCN for the final study visit, which will collect the same measures as Visit 8. Wait-list controls will then be offered the PPLP (Intervention, 3 month Assessment, Follow-up and 6 Month Assessment).
6. Chart review: Participant health care records will be accessed to obtain information on HgA1C and lipid panel tests done during the period of study (Baseline to 6 month assessment).

Data Entry and Analysis: Changes (pre to post-intervention) in dietary adherence, diabetes self-efficacy, quality of life, weight, BMI, Body composition, BP, HgA1C, high density lipoprotein (HDL), low density lipoprotein (LDL), triglycerides (TG) and cholesterol will be assessed and compared within and between PPLP and CON groups. Patient feedback of health/behaviour outcomes will be provided at the end of the study.

Objective 2) Qualitative study to assess strengths, limitations and satisfaction with approach:

At the 3 month clinic visit, the participants from the PPLP group will participate in a focus group discussion to understand adoption of information gained during intervention and to evaluate the barriers/facilitators to adoption. The investigators will also collect copies of the workbooks from participants for process evaluation, to understand factors influencing program retention, success in meeting goals etc. The HCP will participate in a one-on-one interview sessions at this period. Questions will focus on core RE-AIM domains. Responses will help understand adoption of the program at a system level, implementation relative to efficacy and economic constraints, suggestions for improvement and maintenance of PPLP.

Potential Outcomes and Impact of the Proposed Research:

This study will provide important information about the efficacy and suitability of the PPLP for a PCN-based implementation to manage T2D in people from Alberta. The investigators hypothesize that PPLP participants will have improved nutrition and physical activity-related knowledge and skills to manage T2D resulting in better health. Results from this study will inform the success of the program at an individual and system level. This can be used as evidence to justify further scale and spread of the LI to other PCNs and through programs offered by the Alberta Health Services. Furthermore, PPLP being based on 4-A Framework is adaptable, using PPLP as a template; other jurisdictions may be supported to develop similar programming adapted to their local environment. The PI is currently Scientific Director of the Diabetes, Obesity and Nutrition Strategic Clinical Network of Alberta Health Services (AHS), part of whose mission is to advance evidence-based interventions into care. KT materials, in the form of written, oral and e-briefs will be provided regularly to each PCN site and AHS, to provide early evidence of outcomes in each of the RE-AIM domains. PCN personnel from both sites will share their experiences and learn from each other through ongoing e-meetings. Widespread access to all the tools developed will be made through electronic means (PPEP website), and patient-oriented dissemination through CDA, Alberta Diabetes Institute and other venues

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes, Able to read and write in English

Exclusion Criteria:

* Type 1 Diabetes, having severe gastrointestinal issues or diabetes complications requiring specialized diet

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Hb A1C | Baseline, 3month, 6 month
  Hb A1c will be measured at baseline, after intervention at 3 and 6 months. Changes in the test result pre and post intervention will be calculated

SECONDARY OUTCOMES:
10 Item Perceived Dietary Adherence Questionnaire | Baseline, 3 and 6 months.
  Self reported adherence to dietary recommendations by Canadian Diabetes Association Nutrition Therapy Guidelines and Eating Well with Canada's Food Guide. Each item is scored 0-7(0=poor adherence, 7=maximum adherence) yielding a score of 0-77.
8 item Nutrition Self Efficacy | Baseline, 3 and 6 months.
  Self reported changes in nutrition self efficacy. Each item is scored 1-10 (1=not confident, 10=totally confident) yielding a score of 8-80.
5 Item Quality of Life | Baseline, 3 and 6 months.
  Self reported changes in quality of life. Each item is scored 1-5 (1=extreme difficulty in caring normal activities, 5=no problems)
Physical Activity Questionnaire | Baseline, 3 and 6 months.
  Self reported physical activity. It includes 3 subscales - assessing physical activity at work, leisure and sports.
Pedometer Steps Record | Baseline, 3 and 6 months.
  Participants will record steps taken for consecutive 3 days in a week.
Changes in Lipid Panel Test | Baseline, 3 and 6 months
  LDL, HDL, triglycerides and total cholesterol will be measured at baseline and after intervention at 3 and 6 month study periods. Differences in test outcomes pre and post intervention will be calculated.
Changes in Blood Pressure | Baseline, 3 and 6 months
  Systolic and Diastolic BP will be measured at baseline and after intervention at 3 and 6 month study periods. Differences in test outcomes pre and post intervention will be calculated.
Change in Weight | Baseline, 3 and 6 months.
  Weight will be measured at baseline and after intervention at 3 and 6 months study periods. Difference in weight (baseline to 3 months, 3 months to 6 months and baseline to 6 months ) will be calculated
Height (m) | Baseline
  Height will be measured at the baseline visit.
Changes in BMI(kg/m^2) | Baseline, 3 and 6 months
  BMI will be calculated at baseline, 3 and 6months periods using the formula (kg/m^2). BMI will be calculated using the weight measured at each assessment respectively and the measured height from baseline visit. Difference in BMI (baseline to 3 months, 3 months to 6 months and baseline to 6 months ) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Chan, PI, Principal Investigator — Professor
Locations (1):
- Sherwood Park Primary Care Network, Sherwood Park, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Not anticipated

REFERENCES:
- [Background] Asaad G, Soria-Contreras DC, Bell RC, Chan CB. Effectiveness of a Lifestyle Intervention in Patients with Type 2 Diabetes: The Physical Activity and Nutrition for Diabetes in Alberta (PANDA) Trial. Healthcare (Basel). 2016 Sep 27;4(4):73. doi: 10.3390/healthcare4040073. PMID 27690122
- [Background] Raine KD. Determinants of healthy eating in Canada: an overview and synthesis. Can J Public Health. 2005 Jul-Aug;96 Suppl 3(Suppl 3):S8-14, S8-15. doi: 10.1007/BF03405195. PMID 16042158